CLINICAL TRIAL: NCT02295501
Title: A Prospective, Open Label Observational, Phase 1 Safety Study of Passive Immune Therapy During Acute Ebola Virus Disease Using Transfusion of INTERCEPT Plasma Prepared From Volunteer Donors Who Have Recovered From Ebola Virus Disease
Brief Title: A Prospective, Open Label, Phase 1 Safety Study of Passive Immune Therapy During Acute Ebola Virus Disease Using Transfusion of INTERCEPT Plasma Prepared From Volunteer Donors Who Have Recovered From Ebola Virus Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated on expiry of the frozen and stored plasma components.
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI 00113
Record Dates: First submitted 2014-11-04; First posted 2014-11-20 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Acute Ebola Virus Disease
Keywords: Pathogen inactivation; ebola; convalescent plasma; EBOV; amotosalen; Provide access to the potential therapeutic benefit of EBOV convalescent plasma containing antibodies to EBOV.
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EBOV convalescent donors (Experimental): EBOV convalescent donors for passive immune therapy in subjects with acute EVD
  Interventions: Biological: INTERCEPT Plasma

INTERVENTIONS:
Biological: INTERCEPT Plasma — Plasma will be collected from eligible volunteer donors who have recovered from acute EVD (see EBOV convalescent donor inclusion criteria). This donor plasma will be collected by apheresis donation (approximately 650-1300 mL per donation at physician discretion) and treated with the IBS for plasma.
  Other Names: INTERCEPT Blood System for Plasma

SUMMARY:
The objective of this Phase 1 safety study is to provide access to the potential therapeutic benefit of EBOV convalescent plasma containing antibodies to EBOV. The risk of exposure to plasma from donors who may be infected with other transfusion-transmitted pathogens, not detectable by current licensed donor testing procedures, will be mitigated by using pathogen inactivation to minimize the risk of the TTI from these donors, who would otherwise be deferred and ineligible for blood donation.

DETAILED DESCRIPTION:
The objective of this Phase 1 safety study is to provide access to the potential therapeutic benefit of EBOV convalescent plasma containing antibodies to EBOV. The risk of exposure to plasma from donors who may be infected with other transfusion-transmitted pathogens, not detectable by current licensed donor testing procedures, will be mitigated by using pathogen inactivation to minimize the risk of the TTI from these donors, who would otherwise be deferred and ineligible for blood donation.

The study is designed as a prospective, open label, multi-center, single arm study to evaluate the safety and efficacy of INTERCEPT plasma prepared from EBOV convalescent donors for passive immune therapy in subjects with acute EVD.

Data will be collected to assess the safety of this intervention by monitoring adverse events in the immediate 24-hour post transfusion period. Efficacy will be assessed by monitoring the clinical status of treated subjects with respect to clearance of EBOV by using nucleic acid assays to measure pre and post treatment viral titers. A number of clinical parameters indicative of end-organ damage during acute EVD will be monitored to determine if passive immune therapy affects the onset and duration of renal failure and acute lung injury. In addition, blood samples will be collected pre and post transfusion of convalescent EBOV INTERCEPT plasma to determine if biomarkers of endothelial injury are impacted, and if they can be used to guide plasma transfusion therapy to establish a dosing regimen and duration of treatment.

ELIGIBILITY:
Inclusion Criteria:

EBOV Convalescent Donor Inclusion Criteria:

* Recovered from Ebola Virus Disease (EVD) by clinical criteria and declared clinically asymptomatic of active EVD.
* Twenty-eight (28) days from hospital discharge.
* Two negative test results for EBOV nucleic acid by a sensitive nucleic acid test method with blood samples drawn at least 48 hours apart.
* Plasma/serum tested for HIV, HTLV, HCV, HBV, syphilis, and other pathogens (per institutional practice) using licensed test methods. Inclusion of donors with positive test results for these pathogens will be at the discretion of treating physicians, with respect to the relative benefit of donor subject convalescent plasma treated with INTERCEPT pathogen inactivation, compared to the risk to recipients of not receiving EBOV convalescent plasma transfusion therapy.
* ABO blood group and RhD typing performed and donor anti-A and anti-B titers performed.
* Plasma/serum tested for human leukocyte antigen (HLA) antibodies for female donors with history of pregnancy and for donors with a history of transfusions (per institutional practice) using licensed test methods for transfusion-related acute lung injury (TRALI) risk mitigation. Inclusion of donors with positive test results will be at the discretion of treating physicians, with respect to the relative benefit of donor subject convalescent plasma compared to the risk to recipients of not receiving EBOV convalescent plasma transfusion therapy.
* Measurement of antibodies to EBOV, when feasible and ultimately measurement of neutralizing antibodies to EBOV, when available.
* Conformity to age and weight standards for blood donors for plasma donation. Variance from standards may be acceptable with evaluation by treating physician(s) and with donor or legal guardian consent for non-conforming donors when collection of reduced volumes of plasma may be of therapeutic value.
* Cleared by treating physician for apheresis plasma donation.
* Written signed informed consent to donate 650-1300 mL plasma by apheresis at frequencies of twice per week, at the discretion of the treating physician.

Recipient Subject Inclusion Criteria:

* Acute EVD diagnosed by nucleic acid testing and meeting established case definitions (World Health Organization 2014).
* Subject or legal guardian provides written informed consent to receive INTERCEPT plasma.

Exclusion Criteria:

EBOV Convalescent Donor Exclusion Criteria:

• Active EVD

Recipient Subject Exclusion Criteria:

• Documented food allergy to psoralens

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-12; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who survive EVD | through hospital discharge up to 1 year
Proportion of subjects with adverse events | Up to 24 hours post transfusion
Proportion of subjects with Serious Adverse Events | Up to 7 days post-transfusion

SECONDARY OUTCOMES:
Time from diagnosis of acute EVD to death due to acute EVD | censored at hospital discharge up to 1 year
Proportion of subjects with clinical remission, where clinical remission is defined as absence of clinical symptoms indicative of EVD and at least two negative EBOV nucleic acid tests at least 48 hours apart prior to hospital discharge. | through hospital discharge up to 1 year
Time from diagnosis of acute EVD to clinical remission. | through hospital discharge up to 1 year
Reduction of EBOV viral load titers by nucleic acid testing prior to hospital discharge. | through hospital discharge up to 1 year
Subject hemostatic function pre INTERCEPT plasma and post last INTERCEPT plasma transfusion (prior to discharge), as available: o Prothrombin time o International Normalized Ratio (INR) o Activated partial thromboplastin time o Fibrinogen activity | pre and post transfusion up to 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - University of Nebraska Medical Center, Omaha, Nebraska

REFERENCES:
- [Result] Dean CL, Hooper JW, Dye JM, Zak SE, Koepsell SA, Corash L, Benjamin RJ, Kwilas S, Bonds S, Winkler AM, Kraft CS. Characterization of Ebola convalescent plasma donor immune response and psoralen treated plasma in the United States. Transfusion. 2020 May;60(5):1024-1031. doi: 10.1111/trf.15739. Epub 2020 Mar 4. PMID 32129478